CLINICAL TRIAL: NCT06419530
Title: A Double-blind Randomized Clinical Trail Study on the Effectiveness and Safety of Probiotic Formula in Autistic Children With Gastrointestinal Symptoms
Brief Title: A Study on Probiotic Formula in Autistic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Associate director / Associate professor, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMMU-DP-ASD-PMT-20240510
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Gut microbiota
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): In this arm, 4 placebo capsules would be oral administered by participants everyday for 84 days.
  Interventions: Other: placebo capsule
- Fecal microbiota transplantation (FMT) group (Active Comparator): In this arm, 4 FMT capsules would be oral administered by participants everyday for 84 days.
  Interventions: Other: FMT capsule
- Probiotic formula group (Experimental): In this arm, 4 Probiotic formula capsules would be oral administered by participants everyday for 84 days.
  Interventions: Other: Probiotic formula capsule

INTERVENTIONS:
Other: Probiotic formula capsule — The subjects take 4 capsules a day for 84 days.
  Arms: Probiotic formula group
Other: placebo capsule — The subjects take 4 capsules a day for 84 days.
  Arms: Placebo group
Other: FMT capsule — The subjects take 4 capsules a day for 84 days.
  Arms: Fecal microbiota transplantation (FMT) group

SUMMARY:
A Randomized controlled double-blind clinical study on the effectiveness and safety of probiotic formula in Autistic children with gastrointestinal symptoms.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder of children with estimated prevalence of near 1% by WHO in 2022. To date, the cause and etiology of ASD is still unknown, and there is no proven effective pharmacological treatment for ASD. The gut microbiota has been proved to have great impact on neurological development, in this study, we aim to explore the effectiveness of safety of probiotic formula on ASD children, by comparing with placebo and fecal microbiota transplantation (FMT). This study will be a randomized, double-blind, placebo-controlled trial. Totally, 156 Autistic children with gastrointestinal symptoms will be enrolled and randomly allocated into three groups: probiotic formula group, fecal microbiota transplantation (FMT) group and placebo group. participants are treated with 4 probiotic formula/FMT/placebo capsules each day, for 84 days. Participants would be followed up at the 4th, 8th, 12th and 24th week after enrollment by simple physical examination, relevant scale questionaire (including Autism Behavior Checklist(ABC),Childhood Autism Rating Scale(CARS),Gastrointestinal Symptom Rating Scale(GSRS),Social Responsiveness Scale(SRS),Self-Rating Anxiety Scale(SAS) and Autism Diagnostic Observation Schedule(ADOS)), and blood and fecal samples collection.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 3-11 years old
* Clinical diagnosis of ASD, based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* Associated with gastrointestinal symptoms for at least 14 days (diarrhea, constipation, abdominal pain, bloating and/or food allergies/intolerances)
* With guardians who can fully understand the informed consent and voluntarily sign the written informed consent

Exclusion Criteria:

* Antibiotics or probiotics used within 1 mont
* Serious gastrointestinal problems that require immediate treatment (such as life-threatening intestinal obstruction, intestinal perforation, intestinal bleeding
* Medications related to mental disorders or depression
* Relying on tube feeding
* Swallowing dysfunction that unable to take capsules
* History of severe allergies
* Paticipation in other clinical studies within 4 weeks
* Poor compliance and have difficulty in completing follow-up.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Behavioral Rating Scale (ABC) scores of children with autism in 12th week and baseline | week 12
  This scale lists 57 items of abnormal performance in sensation, behavior, emotion and language, and makes the judgment of "yes" and "no" in each item. (the informant refers to the parents of the child or those who have lived with the child for more than two weeks.) when scoring, make "yes" and "no" to each item, "yes" is the symbol"√", and "no" is not marked. The total score of "yes" items is 158, and the screening limit is 53-67 points. 53 points were used as the diagnostic threshold of autism, and the diagnosis score was 67 points.

SECONDARY OUTCOMES:
Changes in Childhood Autism Rating Scale(CARS) before and after treatment | week 0,4,8,12,24
  The scale consists of 15 items, which are used by the examiners. Each item of the scale was scored according to 1-4 grades. The total score was greater than or equal to 30 points for diagnosis of autism, less than 36 points for mild-moderate autism, and for severe autism when the total score reached or greater than 36 points.
Changes in Social Responsiveness Scale(SRS) before and after treatment | week 0,4,8,12
  The scale is composed of 65 items in 5 subscales. The content of the scale mainly involves children's daily social situations, including social perception, cognition, communication, motivation, autistic behavior and other aspects. The scale adopts a 4-point rating, and each item has four options: never, sometimes, often, and always, and is completed by parents or long-term caregivers. The higher the score, the more severe the social impairment and autistic behavior.
Changes in Self-Rating Anxiety Scale(SAS) before and after treatment | week 0,4,8,12
  The scale consists of 20 items. Each item is scored on a scale of 1 to 4, and the final score is the sum of the scores for the 20 items. The final score is multiplied by 1.25 to obtain the integer part, and the standard score is obtained. An anxiety total score below 50 is considered normal; 50-60 is mild, 61-70 is moderate, and above 70 is severe anxiety.
Changes in Autism Diagnostic Observation Schedule(ADOS) before and after treatment | week 0,4,8,12
  The scale is a semi-structured, standardized assessment that includes communication, social interaction, play, and restrictive and repetitive behaviors.
Changes in Gastrointestinal Symptom Rating Scale(GSRS) before and after treatment | week 0,4,8,12, 24
  The scale is a tool commonly used to measure gastrointestinal symptoms. It contains multiple dimensions and items to evaluate the patient's gastrointestinal health status through scoring.
Changes in Serum neurotransmitters (5-HT、GABA、Dopamine) of children with autism before and after treatment | week 0,12
  There are abnormal changes in erum neurotransmitters (including 5-HT, GABA, and dopamine) in autistic children.In order to explore whether "Precision Microbiota Transplantation" can improve serum neurotransmitters (including 5-HT, GABA, and dopamine) levels.
Changes in gut microbiota of children with autism before and after treatment | week 0,12
  There are abnormal changes in intestinal flora in autistic children.In order to explore whether "Precision Microbiota Transplantation" can improve the level of intestinal flora.
Changes in Behavioral Rating Scale (ABC) scores of children with autism before and after treatment | week 0,4,8, 24
  This scale lists 57 items of abnormal performance in sensation, behavior, emotion and language, and makes the judgment of "yes" and "no" in each item. (the informant refers to the parents of the child or those who have lived with the child for more than two weeks.) when scoring, make "yes" and "no" to each item, "yes" is the symbol"√", and "no" is not marked. The total score of "yes" items is 158, and the screening limit is 53-67 points. 53 points were used as the diagnostic threshold of autism, and the diagnosis score was 67 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei, MD, Principal Investigator — Daping Hospital,Army medical university
Locations (1):
- Department of Gastroenterology, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China